CLINICAL TRIAL: NCT01462669
Title: An Open-label, Randomized, Single Centre, 4-way Crossover Study to Evaluate the Pharmacokinetics of Single Oral Doses of Ezogabine/Retigabine in Healthy Adult Taiwanese Subjects
Brief Title: Crossover Study to Evaluate the Pharmacokinetics of Ezogabine/Retigabine in Taiwanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 115860
Record Dates: First submitted 2011-10-27; First posted 2011-10-31 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Epilepsy
Keywords: Ezogabine; Pharmacokinetics; Retigabine
MeSH Terms: conditions — Epilepsy | interventions — ezogabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Period 1 (Other): A single 50mg ezogabine/retigabine tablet will be administered orally with the subject in the fasted state
  Interventions: Drug: 50mg Ezogabine/retigabine
- Treatment Period 2 (Other): A single 100mg ezogabine/retigabine tablet will be administered orally with the subject in the fasted state
  Interventions: Drug: 100mg Ezogabine/retigabine
- Treatment Period 3 (Other): A single 200mg ezogabine/retigabine tablet will be administered orally with the subject in the fasted state
  Interventions: Drug: 200mg Ezogabine/retigabine
- Treatment Period 4 (Other): A single 400mg ezogabine/retigabine tablet will be administered orally with the subject in the fasted state
  Interventions: Drug: 400mg Ezogabine/retigabine

INTERVENTIONS:
Drug: 50mg Ezogabine/retigabine — A single 50mg ezogabine/retigabine tablet will be administered orally with the subject in the fasted state
  Other Names: GW582892
  Arms: Treatment Period 1
Drug: 100mg Ezogabine/retigabine — A single 100mg ezogabine/retigabine tablet will be administered orally with the subject in the fasted state
  Other Names: GW582892
  Arms: Treatment Period 2
Drug: 200mg Ezogabine/retigabine — A single 200mg ezogabine/retigabine tablet will be administered orally with the subject in the fasted state
  Other Names: GW582892
  Arms: Treatment Period 3
Drug: 400mg Ezogabine/retigabine — A single 400mg ezogabine/retigabine tablet will be administered orally with the subject in the fasted state
  Other Names: GW582892
  Arms: Treatment Period 4

SUMMARY:
The purpose of this study is to investigate the pharmacokinetics of single oral doses of ezogabine/retigabine and the primary metabolite (NAMR) in healthy male and female Taiwanese volunteers. Subjects will receive four separate doses of ezogabine/retigabine tablets: 50 mg, 100 mg, 200 mg and 400 mg administered once orally. Blood samples will be obtained at pre-defined timepoints over the duration of the study to determine the concentration of ezogabine/retigabine and NAMR. Safety assessments will include measurements of vital signs, collection of adverse events, clinical laboratory tests and the Columbia Suicide Severity Rating Scale.

DETAILED DESCRIPTION:
Ezogabine/retigabine (GW582892), N-[2-amino-4(4-fluorobenzylamino)-phenyl] carbamic acid ethyl ester, is a novel anti-epileptic compound which has been developed as an adjunctive treatment for partial onset seizures in patients with refractory epilepsy.

This is an open-label, randomized, single-center, 4-way crossover study to investigate the pharmacokinetics of single oral doses of ezogabine/retigabine and the n-acetyl metabolite of ezogabine/retigabine (NAMR) in healthy male and female Taiwanese volunteers. The study consists of a screening phase, 4 treatment periods and a follow-up visit. Subjects will receive each of the following four treatments administered in a randomized four-way crossover design: 50 mg, 100 mg, 200 mg and 400 mg ezogabine/retigabine tablets administered once orally. Serial blood samples will be obtained at pre-defined timepoints for pharmacokinetic analysis of ezogabine/retigabine and NAMR. Safety assessments will include measurements of vital signs, collection of adverse events, clinical laboratory tests and the Columbia Suicide Severity Rating Scale.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Male or female between 20 and 65 years of age inclusive, at the time of signing the informed consent.
2. Taiwanese ancestry defined as being born in Taiwan, having four ethnic Chinese/Taiwanese grandparents, holding a Taiwanese passport or identity papers and subject is able to speak Chinese/Taiwanese.
3. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and 12-lead ECG. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
4. Body weight ≥ 50 kg and BMI within the range 18.5-24.9 kg/m2 (inclusive).
5. A female subject is eligible to participate if she is of:

   * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol <40 pg/ml (<147 pmol/L) is confirmatory]. Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the contraception methods in Section 8.1 if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrollment. For most forms of HRT, at least 2-4 weeks will elapse between the cessation of therapy and the blood draw; this interval depends on the type and dosage of HRT. Following confirmation of their post-menopausal status, they can resume use of HRT during the study without use of a contraceptive method.
   * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 1 week post-last dose of GW582892.
6. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
7. AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
8. Normal ECG morphology and measurements. In particular QTcB or QTcF < 450 msec or QTc < 480 msec in subjects with Bundle Branch Block based on an average from three ECGs obtained over a brief recording period.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

1. Subject has made a suicide attempt in the past or, in the investigator's judgment, poses a significant suicide risk. Evidence of serious suicide risk may include any history of suicidal behavior in the past 6 months and/or any suicidal ideation of type 4 or 5 on the Columbia Suicide Severity Rating Scale (C-SSRS).
2. A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening
3. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
4. A positive pre-study drug/alcohol screen.
5. A positive test for HIV antibody.
6. History of regular alcohol consumption within 6 months of the study defined as:

   - An average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 360 ml of beer, 150 ml of table wine or 45 ml of 80 proof distilled spirits.
7. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
8. Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
9. Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study assessments or compromise subject safety.
10. History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
11. Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
12. Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
13. Lactating females.
14. Unwillingness or inability to follow the procedures outlined in the protocol.
15. Subject is mentally or legally incapacitated.
16. History of sensitivity to heparin or heparin-induced thrombocytopenia.
17. Subjects who have asthma or a history of asthma.
18. Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
19. Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pummelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2012-04-10 (Actual); Primary Completion 2012-06-27 (Actual); Study Completion 2012-06-27 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of single oral doses of ezogabine/retigabine and NAMR over the range of 50mg to 400mg in healthy male and female Taiwanese volunteers | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 14 weeks
  Peak plasma concentration (Cmax) of ezogabine/retigabine; and area under the plasma concentration-time curve from time zero to infinity (AUC(0-∞)) for ezogabine/retigabine

SECONDARY OUTCOMES:
Pharmacokinetics of single oral doses of ezogabine/retigabine and NAMR over the range of 50mg to 400mg in healthy male and female Taiwanese volunteers | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 14 weeks
  Time to peak plasma concentration (Tmax) of ezogabine/retigabine; Terminal phase half-life (t½) of ezogabine/retigabine; Cmax of NAMR; AUC(0-∞) for NAMR; and Tmax of NAMR
Safety and tolerability data after single oral doses of ezogabine/retigabine in healthy male and female Taiwanese volunteers | Participants will be followed and monitored for the duration of their hospital stay. The longest duration of participation in the study will be approximately 14 weeks
  Safety and tolerability data as measured by adverse events, vital signs, ECGs, clinical laboratory measurements and C-SSRS

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Results for study 115860 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/115860?search=study&study_ids=115860#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 115860 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115860 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115860 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115860 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115860 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115860 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 115860 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register